CLINICAL TRIAL: NCT04686916
Title: A Randomised, Double-Blind, Placebo-Controlled, Crossover Trial Studying the Efficacy and Safety of IP2018 in Young, Depressed, Erectile Dysfunction (ED) Patients
Brief Title: Clinical Trial Studying the Efficacy and Safety of IP2018 in Depressed, Erectile Dysfunction (ED) Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Initiator Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IP2018CS01
Record Dates: First submitted 2020-12-09; First posted 2020-12-29 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-08

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IP2018_dose 1 (Experimental): IP2018_dose1
  Interventions: Drug: IP2018
- IP2018_dose 2 (Experimental): IP2018_dose2
  Interventions: Drug: IP2018
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IP2018 — Test drug
  Arms: IP2018_dose 1; IP2018_dose 2
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase IIa, randomised, double-blind, placebo-controlled, 3-period, crossover study to assess two single oral dose levels of IP2018. It is planned to enrol 24 patients. Patients will take part in three treatment periods, in which they will be randomised to receive either a single dose of IP2018 or a single dose of placebo in each treatment period.

ELIGIBILITY:
Inclusion Criteria:

- Male patients with a diagnosis of mild to moderate depression and ED as determined from the Hamilton depression scale score of 7 to 23 and International Index of Erectile Function (IIEF-5) score of 12 to 18, respectively, with a body mass index of 18 to 32 kg/m2 (inclusive), of any ethnic origin.

Exclusion Criteria:

- Any significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal (GI), haematological, endocrinological, metabolic, neurological, psychiatric conditions, or history of fainting or syncope or such condition that, in the opinion of Investigator, may place the patient at unacceptable risk as a participant in the study, may interfere with the interpretation of safety or tolerability data obtained in this study, or may interfere with the absorption, distribution, metabolism or excretion of drugs, or with the completion of treatment according to this protocol.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male patients with a diagnosis of mild to moderate depression and erectile dysfunction
Enrollment: 24 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Erectile Function | A 6 hours time interval after dosing
  Rigiscan device assessment of tumescence

SECONDARY OUTCOMES:
Safety assessment | From randomisation to end of study participation
  Clinical safety data from AE reporting, 12-lead electrocardiograms (ECGs), vital signs (standing and supine blood pressure, heart rate and oral temperature [supine only]), physical examinations and clinical laboratory evaluations
Pharmacokinetics of IP2018 | From start to end of assessments
  AUC
Pharmacokinetics of IP2018 | From start to end of assessment
  Tmax

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Fiore Fiore, MD, Principal Investigator — MAC UK
Locations (1):
- MAC, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No